CLINICAL TRIAL: NCT03926650
Title: Correlation of Train Of Four (TOF) With Frontal EMG Parameter Measured by Patient State Index (PSI) Monitor in Extubation Phase of General Anesthesia
Brief Title: The Correlation Between the Frontal Electromyography Parameter in Patient State Index (PSI) Monitor and Train of Four
Status: Completed | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Hakan Gokalp TAS, Research Assistant Doctor Hakan Gökalp TAŞ, Erzincan University
Other Study IDs: ErzincanUnv
Record Dates: First submitted 2019-04-18; First posted 2019-04-24 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Masimo Sedline Monitor Patient State Index — Masimo Sedline Monitor shows frontal electromyography and patient state index, Train of four monitor shows muscle strength on adductor pollicis muscle
  Other Names: Train Of Four

SUMMARY:
The Train Of Four (TOF) Monitor will be placed on ulnar nerve on right wrist of the patients who has surgery under general anaesthesia. This is for stimulation of adductor pollicis muscle. Sedline (Masimo Electromyography(EMG) and Patient State Index(PSI)) Monitor will be placed on the frontal area of head. After the induction of general anaesthesia the investigators will wait for disappearance of eyelash reflex. TOF monitor will be calibrated and muscle relaxant will be applied. After TOF is %0 and disappearance of thumb movement the patient will be intubated. After surgery the investigators will apply muscle relaxant reversal drugs. Then the investigators will record PSI and EMG parameters when TOF is %0, %25, %50,%75,%90. When TOF is %90 the investigators will extubate the patient. The investigators will record PSI and EMG parameters after 5 minutes.

DETAILED DESCRIPTION:
The study is planned prospective and observational. The study started after approval of Erzincan Binali Yıldırım University Ethics Committee and taking written approval of patients. The study includes 84 patients who has surgery continues more then 1 hour, who is between ages 18-65, who is ASA I,II and III. The patients who has allergical reactions of the drugs used, neurological or neuromuscular diseases,the patients who use drugs effecting the neuromuscular junction, pregnant patients, electrolyte disregulations, major organ failures, liver failure, kidney failure, obese and cachectic patients are excluded from the study.

All patients will be informed and signed written approval 1 day before the surgery. Patients will be taken to the operating room, venous catheter will be applied on antecubital area. 3 channel EKG , SpO2 Monitor and noninvasive blood pressure monitorisation will be applied. The patients will be taken 2-4 litres of O2 with nasal cannula .The Train Of Four (TOF) Monitor will be placed on ulnar nerve on right wrist of the patients who has surgery under general anaesthesia. This is for stimulation of adductor pollicis muscle. Sedline (Masimo Electromyography(EMG) and Patient State Index(PSI)) Monitor will be placed on the frontal area of head. After the induction of general anaesthesia the investigators will wait for disappearance of eyelash reflex. TOF monitor will be calibrated and muscle relaxant will be applied. After TOF is %0 and disappearance of thumb movement the patient will be intubated. After surgery the investigators will apply muscle relaxant reversal drugs. PSI and EMG parameters will be recorded when TOF is %0, %25, %50,%75,%90. When TOF is %90 the investigators will extubate the patient. PSI and EMG parameters will be recorded after 5 minutes. The patient will be taken to the PACU room. On 5,10,30 minutes after surgery, the investigators will record aldrete score of patients.

ELIGIBILITY:
Inclusion Criteria:

* surgery continues more then 1 hour
* between ages 18-65
* ASA I,II and III patients

Exclusion Criteria:

* The patients who has allergical reactions of the drugs used
* neurological or neuromuscular diseases
* the patients who use drugs effecting the neuromuscular junction
* pregnant patients
* electrolyte disregulations
* major organ failures, liver failure, kidney failure
* obese and cachectic patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients wha has surgery continues more then 1 hour
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Patient State Index | 0 minutes
  Measures anaesthetic awakeness. It can be between 0-100. The investigators will record this parameter after using the reversal drugs
Patient State Index | 1 minutes
  Measures anaesthetic awakeness. It can be between 0-100. The investigators will record this parameter after using the reversal drugs
Patient State Index | 2 minutes
  Measures anaesthetic awakeness. It can be between 0-100. The investigators will record this parameter after using the reversal drugs
Patient State Index | 3 minutes
  Measures anaesthetic awakeness. It can be between 0-100. The investigators will record this parameter after using the reversal drugs
Patient State Index | 4 minutes
  Measures anaesthetic awakeness. It can be between 0-100. The investigators will record this parameter after using the reversal drugs
Patient State Index | 5 minutes
  Measures anaesthetic awakeness. It can be between 0-100. The investigators will record this parameter after using the reversal drugs
Electromyography (Frontal EMG) | 0 minutes
  Measures frontal muscles' strength.It can be between % 0 - %100. The investigators will record this parameter after using the reversal drugs
Electromyography (Frontal EMG) | 1 minutes
  Measures frontal muscles' strength.It can be between % 0 - %100. The investigators will record this parameter after using the reversal drugs
Electromyography (Frontal EMG) | 2 minutes
  Measures frontal muscles' strength.It can be between % 0 - %100. The investigators will record this parameter after using the reversal drugs
Electromyography (Frontal EMG) | 3 minutes
  Measures frontal muscles' strength.It can be between % 0 - %100. The investigators will record this parameter after using the reversal drugs
Electromyography (Frontal EMG) | 4 minutes
  Measures frontal muscles' strength.It can be between % 0 - %100. The investigators will record this parameter after using the reversal drugs
Electromyography (Frontal EMG) | 5 minutes
  Measures frontal muscles' strength.It can be between % 0 - %100. The investigators will record this parameter after using the reversal drugs

CONTACTS AND LOCATIONS:
Overall Officials: Hakan G. Taş, Principal Investigator — Mengucek Gazi Education and Research Hospital
Locations (1):
- Erzincan University, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No